CLINICAL TRIAL: NCT02645240
Title: Predictive Factors of Intestinal Infraction in Patients With Acute Mesenteric Ischemia
Brief Title: Predictive Factors of Intestinal Infraction in Acute Mesenteric Ischemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: mansoura30
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Mesenteric Ischemia
MeSH Terms: conditions — Mesenteric Ischemia | interventions — Heparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Heparin injection (Experimental): Injection of low molecular weight heparin in patients with acute mesenteric ischemia to assess outcome
  Interventions: Drug: Heparin injection

INTERVENTIONS:
Drug: Heparin injection — Intravenous heparin injection in patients with acute mesenteric ischemia and evaluating their response within 24 hours
  Other Names: Low molecular weight heparin injection

SUMMARY:
The study aims to identify several factors that can accurately predict the incident of intestinal infraction in patients with mesenteric vascular occlusion or ischemia.

DETAILED DESCRIPTION:
The study aims to identify several clinical, laboratory, and radiologic factors that can accurately predict the occurrence of intestinal infraction in patients with mesenteric vascular occlusion or ischemia in order to prevent unnecessary surgical intervention in patients with just intestinal ischemia and to hasten intervention in patients with actual intestinal gangrene.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute mesenteric Ischemia

Exclusion Criteria:

* Patients with other causes of acute abdomen other than mesenteric Ischemia

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-10; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 48 hours
  Number of patients with resolved abdominal symptoms and incidence of patients developing shock

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D, Principal Investigator — Mansoura Univesity
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided